CLINICAL TRIAL: NCT03859414
Title: A Single-center, Randomized, Double-blind, Single Dose, 4-way Cross-over, Placebo-controlled Ethnic Sensitivity Study to Assess the Pharmacokinetics (PK), Pharmacodynamics (PD), Safety, and Tolerability of Different Dosages of CHF 5993 Pressurized Metered Dose Inhaler (pMDI) in Caucasian and Japanese Healthy Subjects
Brief Title: PK of BDP/FF/GB Single-inhaler Triple Therapy in Japanese vs. Caucasians
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: CLI-05993AB4-01; 2018-003310-40 (EudraCT Number)
Record Dates: First submitted 2019-02-18; First posted 2019-03-01 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: 4-way Crossover Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Therapeutic Dose 1 (Active Comparator): Single dose administration of CHF 5993 100/6/12.5 µg pMDI 2 inhalations. Total dose of CHF 5993 pMDI = 200/12/25 µg
  Interventions: Drug: Therapeutic Dose 1
- Therapeutic Dose 2 (Active Comparator): Single dose administration of CHF 5993 200/6/12.5 µg pMDI 2 inhalations. Total dose of CHF 5993 pMDI = 400/12/25 µg
  Interventions: Drug: Therapeutic Dose 2
- Supra-therapeutic Dose (Active Comparator): Single dose administration of CHF 5993 100/6/12.5 µg pMDI 8 inhalations Total dose of CHF 5993 pMDI = 800/48/100 µg
  Interventions: Drug: Supra-therapeutic Dose
- Placebo (Placebo Comparator): Single dose administration of CHF 5993 pMDI placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Therapeutic Dose 1 — CHF 5993 100/6/12.5 µg pMDI, fixed combination of BDP 100 µg + FF 6 µg + GB 12.5 µg.
  Arms: Therapeutic Dose 1
Drug: Therapeutic Dose 2 — CHF 5993 200/6/12.5 µg pMDI, fixed combination of BDP 200 µg + FF 6 µg + GB 12.5 µg.
  Arms: Therapeutic Dose 2
Drug: Supra-therapeutic Dose — CHF 5993 200/6/12.5 µg pMDI, fixed combination of BDP 200 µg + FF 6 µg + GB 12.5 µg.
  Arms: Supra-therapeutic Dose
Drug: Placebo — CHF 5993 placebo pMDI
  Arms: Placebo

SUMMARY:
The purpose of conducting this study is to obtain PK data of Beclometasone Dipropionate (BDP)/Beclometasone-17-MonoPropionate (B17MP), Formoterol Fumarate (FF) and Glycopyrronium Bromide (GB) after inhalation of CHF 5993 in Japanese as well as Caucasian healthy subjects under the same setting.

DETAILED DESCRIPTION:
The Study is single-centre, randomized, double-blind, single-dose, 4-way cross-over, placebo-controlled.

The safety, tolerability, PD and PK of CHF 5993 will be assessed in Japanese and Caucasian healthy volunteers.

A total of 32 healthy male and female volunteers are planned to be included where they will receive four different treatments (study drug or placebo) over four treatment periods.

Standard safety assessments will be conducted during the study, including safety blood and urine laboratory tests, liver function tests, vital signs, physical examinations, ECGs, 24-hour Holter and observations of any adverse events. Blood samples will also be collected for PK analysis. Blood and urine samples will be collected for pharmacodynamics analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subject's written informed consent obtained prior to any study related procedure;
* Healthy male and female subjects aged 20 to 55 years inclusive;
* For Japanese subjects: must be a Japanese subject who has resided outside Japan for no more than 5 years, born in Japan and holding a Japanese passport, with all 4 grandparents Japanese, as confirmed by interview;
* Subject must be willing and able to adhere to the prohibitions and restrictions specified in this protocol and to comply with the correct use of the devices specified in this protocol;
* Body mass index within the range of 18.0 to 25.0 kg/m2 inclusive;
* Non-smokers or ex-smokers who smoked <5 pack years and stopped smoking >1 year prior to screening;
* Subject must be healthy on the basis of physical examination, medical history, vital signs, and 12 -lead digitised Electrocardiogram (12-lead ECG);
* Vital signs (Blood pressure and body temperature) within normal limits;
* 12-lead ECG considered as normal;
* Lung function measurements within normal limits;
* Women of non-childbearing potential (WONCBP) and women of childbearing potential (WOCBP) fulfilling one of the following criteria: a) WOCBP with fertile male partners: they and/or their partner must be willing to use a highly effective birth control method from the signature of the informed consent and until the follow-up visit or b) WOCBP with non-fertile male partners: (contraception is not required in this case).
* Female subject, except if postmenopausal, must have a negative serum beta-human chorionic gonadotropin at screening and a negative urine pregnancy test at Day -1 prior the first drug administration;
* Subjects must agree not to donate sperm or ova from the time of the first administration of study medication until three months after the end of the systemic exposure of the study drug or until the last follow-up visit, whichever occurs later;
* Males fulfilling one of the following criteria: a) Males with pregnant or non-pregnant WOCBP partners: they must be willing to use male condom from the signature of the informed consent and until the follow-up visit or b) Non-fertile male subjects (contraception is not required in this case) or c) Males with partner not of childbearing potential (contraception is not required in this case).

Exclusion Criteria:

* Participation in another clinical trial with an investigational drug in the 90 days or 5 half-lives of non-biological entities of that investigational drug (whichever is longer) preceding the administration of the study drug;
* Clinically relevant and uncontrolled respiratory, cardiac, hepatic, gastrointestinal, renal, endocrine, metabolic, neurologic, or psychiatric disorders that may interfere with successful completion of this study;
* Any other abnormal findings on vital signs, ECG, physical examination or laboratory evaluation of blood and urine samples that the investigator judges as likely to interfere with the study or pose an additional risk in participating;
* Medical diagnosis of narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that in the opinion of the investigator would prevent use of anticholinergic;
* History of asthma, including childhood asthma, Chronic Obstructive Pulmonary Disease (COPD) or any other chronic pulmonary diseases or condition;
* Positive HIV1 or HIV2 serology;
* results from the Hepatitis serology at screening which indicates acute or chronic Hepatitis (i.e. positive HB surface antigen (HBsAg), HB core antibody (anti-HBc), or Hepatitis C (positive HCV antibody);
* Blood donation or blood loss (equal or more than 450 mL), less than 2 months prior to randomisation;
* Abnormal haemoglobin level defined as <12.0 g/dL in females and <14.0 g/dL in males;
* Positive urine test for cotinine at screening or prior to randomisation;
* Unsuitable veins for repeated venepuncture;
* History or clinical evidence of drug and/or alcohol abuse within 12 months prior to screening and randomisation;
* Known intolerance/hypersensitivity to any of the excipients/components contained in any of the formulations used in the trial;
* Taking any drug treatment, including prescribed or Over the Counter (OTC) medicines as well as homeopathic remedies etc., in the 14 days before the screening and prior randomisation, with the exception of occasional paracetamol (maximum 3 g per day with a maximum of 10 g per 14 days for mild non-exclusionary conditions), hormonal contraceptives; hormonal replacement treatment for post-menopausal women, occasional ibuprofen (maximum 1.2 g per day, not to exceed 12 g in the 14 days before the screening);
* Taking enzyme-inducing drugs, enzyme-inhibiting drugs, biologic drugs or any drug known to have a well-defined potential for hepatotoxicity (e.g. isoniazide, nimesulide, ketoconazole) in the 3 months before screening or prior to randomisation;
* Heavy caffeine drinker >28 cups/week of coffee or similar caffeinated beverages e.g., tea, cola per day);
* Bacterial or viral respiratory tract, sinus or middle ear infection affecting health status within 4 weeks prior to randomisation;
* Night shift workers with night shifts within 8 weeks prior to randomisation and during the study.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) of B17MP, formoterol and GB | Over 24 hours after administration for B17MP and FF, over 48 hours after administration for GB
  Area under the plasma concentration versus time curve after a single-dose administration of CHF 5993 pMDI
Maximum of Concentration (Cmax) of B17MP, FF and GB | Over 24 hours after administration for B17MP and FF, over 48 hours after administration for GB
  Peak Plasma Concentration after a single-dose administration of CHF 5993 pMDI

SECONDARY OUTCOMES:
Number of Adverse Events (AEs) | through study completion, an average of 13 weeks
  Assessment of the general safety and tolerability in terms of number of Treatment Emergent Adverse Event (TEAEs), Adverse Drug Reaction (ADRs), serious TEAEs, severe TEAEs and TEAEs leading to study discontinuation and to death.
Number of subjects with Adverse Events | through study completion, an average of 13 weeks
  Assessment of the general safety and tolerability in terms number of subjects with TEAEs, ADRs, serious TEAEs, severe TEAEs and TEAEs leading to study discontinuation and to death.
Percentage of subjects with Adverse Events | through study completion, an average of 13 weeks
  Assessment of the general safety and tolerability in terms of incidence of TEAEs, ADRs, serious TEAEs, severe TEAEs and TEAEs leading to study discontinuation and to death.
Clinical laboratory parameters (biochemistry) | Over 24 hours after administration
  Assessment of PD profile in terms of plasma cortisol, serum potassium and serum glucose after a single-dose administration of CHF 5993 pMDI
Clinical laboratory parameters (urinalysis) | Over 24 hours after administration
  Assessment of PD profile in terms of urine cortisol and creatinine excretion after a single-dose administration of CHF 5993 pMDI
Heart rate | Over 24 hours after administration
  Assessment of PD profile in terms of the Heart Rate after a single-dose administration of CHF 5993 pMDI
12-lead ECG parameters | Over 24 hours after administration
  Assessment of pharmacodynamics profile in terms of 12-lead ECG parameters extracted from Holter after a single-dose administration of CHF 5993 pMDI
Vital signs | Over 24 hours after administration
  Assessment of pharmacodynamics profile in terms of vital signs (systolic and diastolic blood pressure) after a single-dose administration of CHF 5993 pMDI

CONTACTS AND LOCATIONS:
Locations (1):
- Richmond Pharmacology Ltd, London, Tooting, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cella M, Taubel J, Delestre-Levai I, Tulard A, Vele A, Georges G. Ethnic Sensitivity Study of the Extrafine, Single-Inhaler, Triple Therapy Beclomethasone Dipropionate, Formoterol Fumarate, and Glycopyrronium Bromide Pressurized Metered Dose Inhaler in Japanese and Caucasian Healthy Individuals: A Randomized, Double-Blind, Single-Dose Crossover Study. Clin Ther. 2021 Nov;43(11):1934-1947.e4. doi: 10.1016/j.clinthera.2021.09.001. Epub 2021 Sep 29. PMID 34600734